CLINICAL TRIAL: NCT05018221
Title: Better Evidence and Translation for Calciphylaxis
Acronym: BEAT-Calci
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Australasian Kidney Trials Network (Network); Northern Care Alliance NHS Foundation Trust (Other); Waitemata District Health Board (Other Government); Vantive Health LLC (Industry); Berry Consultants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEAT-Calci
Record Dates: First submitted 2021-08-09; First posted 2021-08-24 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Calciphylaxis
MeSH Terms: conditions — Calciphylaxis | interventions — Vitamin K 1; magnesium citrate; sodium thiosulfate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Adaptive, platform, randomized controlled trial, involving multiple interventions spanning several domains of therapeutic care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding of all parties will not be possible for all domains. The default position of the BEAT-Calci platform is that treatments determined by randomization will be blinded to as high a level is feasible.
  Within practical domains, a blind will be adopted, whereby participants, site personnel, trial investigators and outcome assessors will remain blinded to the treatment from the time of randomization until database lock of the comparisons to which that participant is contributing data. In blinded domains, randomization data will not be accessible by anyone else involved in the trial with the following exceptions: (1) data managers who work on the randomization and drug management system, (2) unblinded statistician(s) involved with the response adaptive randomization, and (3) the unblinded biostatistician who prepares reports for the IDMC. Information on the blind, or lack thereof, per domain will be described in the respective Domain-Specific Appendix.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Placebo (Double-Blind Period) (Placebo Comparator): Placebo Vitamin K1 Placebo Magnesium Citrate Placebo Sodium Thiosulphate
  Interventions: Drug: Placebo injection (normal saline); Drug: Placebo capsule (Vitamin K1); Drug: Placebo tablet (Magnesium citrate)
- Vitamin K1 (Double-Blind Period) (Experimental): Dose: 10mg Vitamin K1 capsules, administered 3 times per week following the subject's hemodialysis session.
  * Placebo Magnesium Citrate
  * Placebo Sodium Thiosulphate
  Interventions: Drug: Vitamin K1; Drug: Placebo injection (normal saline); Drug: Placebo tablet (Magnesium citrate)
- Magnesium Citrate (Double-Blind Period) (Experimental): Dose: 150mg Magnesium Citrate tablets, administered 3 times per day. On dialysis days, administration of the middle daily dose should occur following the subject's hemodialysis session.
  * Placebo Vitamin K1
  * Placebo Sodium Thiosulphate
  Interventions: Drug: Magnesium citrate; Drug: Placebo injection (normal saline); Drug: Placebo capsule (Vitamin K1)
- Sodium Thiosulfate (Double-Blind Period) (Experimental): Dose: 25g Sodium Thiosulfate injection, administered intravenously 3 times per week, during the subject's last hour of hemodialysis.
  * Placebo Vitamin K1
  * Placebo Magnesium Citrate
  Interventions: Drug: Sodium Thiosulfate; Drug: Placebo capsule (Vitamin K1); Drug: Placebo tablet (Magnesium citrate)
- High Flux Hemodialysis (Active Comparator): Hemodialysis using a high flux dialyser
  Interventions: Device: High Flux Dialyser
- Medium Cut-off Hemodialysis (Experimental): Hemodialysis using a medium cut-off dialyser
  Interventions: Device: Medium Cut-off Dialyser

INTERVENTIONS:
Drug: Vitamin K1 — Vitamin K1 capsule (10mg) to be administered 3 times per week following the subject's hemodialysis session.
  Other Names: Phytonadione
  Arms: Vitamin K1 (Double-Blind Period)
Drug: Magnesium citrate — Magnesium Citrate tablet (150mg) to be administered 3 times per per day. On dialysis days, administration of the middle daily dose should occur following the subject's hemodialysis session.
  Arms: Magnesium Citrate (Double-Blind Period)
Drug: Sodium Thiosulfate — Sodium Thiosulfate injection (25g/100ml) to be administered intravenously 3 times per week, during the subject's last hour of hemodialysis.
  Other Names: Intravenous Sodium Thiosulfate Injection
  Arms: Sodium Thiosulfate (Double-Blind Period)
Device: High Flux Dialyser — Hemodialysis using a high flux dialyser.
  Other Names: High Flux Hemodialysis
  Arms: High Flux Hemodialysis
Device: Medium Cut-off Dialyser — Hemodialysis using a medium cut-off dialyser.
  Other Names: Medium Cut-off Hemodialysis
  Arms: Medium Cut-off Hemodialysis
Drug: Placebo injection (normal saline) — Placebo to be administered intravenously 3 times per week, during the subject's last hour of hemodialysis.
  Other Names: 0.9% sodium chloride solution
  Arms: Magnesium Citrate (Double-Blind Period); Placebo (Double-Blind Period); Vitamin K1 (Double-Blind Period)
Drug: Placebo capsule (Vitamin K1) — Placebo to be administered 3 times per week following the subject's hemodialysis session.
  Other Names: Matching placebo capsule
  Arms: Magnesium Citrate (Double-Blind Period); Placebo (Double-Blind Period); Sodium Thiosulfate (Double-Blind Period)
Drug: Placebo tablet (Magnesium citrate) — Placebo to be administered 3 times per day. On dialysis days, administration of the middle daily dose should occur following the subject's hemodialysis session.
  Other Names: Matching placebo tablet
  Arms: Placebo (Double-Blind Period); Sodium Thiosulfate (Double-Blind Period); Vitamin K1 (Double-Blind Period)

SUMMARY:
This global platform study will evaluate multiple interventions, across several domains of therapeutic care, in adult patients with kidney failure and newly diagnosed calciphylaxis.

DETAILED DESCRIPTION:
BEAT-Calci is a randomized, adaptive, multi-center, platform trial that will evaluate multiple interventions, across several domains of therapeutic care. The objective of the study is to establish high-quality evidence on the effect of a range of interventions in patients with kidney failure and newly diagnosed calciphylaxis. Calciphylaxis is a rare disease affecting 1-2 people in 10,000.

The trial will commence with a Dialysis Membrane Domain and Pharmacotherapy Domain. The Pharmacotherapy Domain of BEAT-Calci is a placebo-controlled, double blind, response adaptive, randomised controlled trial that will investigate whether any of the pharmacotherapeutic agents is superior to placebo in improving outcomes. The Dialysis Membrane Domain of BEAT-Calci is an open-label, randomised controlled two-way comparison between two different dialysis technologies.

The BEAT-Calci Wound Assessment Scale (BCWAS) is the primary endpoint for the trial. It is an 8-point ordinal categorical scale of disease outcomes and will be used to determine each participant's outcome.

The trial will utilise a Bayesian adaptive sample size re-estimation approach for sample size calculations. The trial will continue to recruit until predefined superiority or futility rules are met. As the trial progresses, in response to information accumulating during the trial, there are various adaptations that can occur, including addition or removal of an intervention arm, response adaptive randomisation and addition of new therapeutic domains.

ELIGIBILITY:
Inclusion Criteria:

1. Currently receiving haemodialysis, or peritoneal dialysis that can be converted to haemodialysis, with planned ongoing haemodialysis a minimum of three times per week for at least the duration of the protocolised calciphylaxis treatments within this trial
2. Have a new calciphylaxis ulcer present for less than 10 weeks
3. Age ≥ 18 years
4. Eligible for randomisation in at least one recruiting domain
5. The participant and treating physician are willing and able to perform trial procedures

Exclusion Criteria:

Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
BEAT-Calci Wound Assessment Scale (BCWAS) - Baseline to Week 12 | Week 12
  To determine whether addition of the intervention changes the sentinel ulcer from Baseline to Week 12 on the BEAT-Calci Wound Assessment Scale. This is an 8-point ordinal categorical scale of change since baseline, which will be used to determine each participant's outcome. The scale is described as:
  1. Complete epithelialisation of the sentinel ulcer
  2. >50% reduction in sentinel ulcer surface area
  3. 20-50% reduction in sentinel ulcer surface area
  4. 0-20% reduction in sentinel ulcer surface area
  5. Any increase in sentinel ulcer surface area
  6. Development of new ulcers
  7. Amputation due to an ulcer
  8. All-cause death

SECONDARY OUTCOMES:
BEAT-Calci Wound Assessment Scale - Baseline to Week 26 | Week 26
  To determine whether addition of the intervention changes the sentinel ulcer from Baseline to Week 26 on the BEAT-Calci Wound Assessment Scale. This is an 8-point ordinal categorical scale of change since baseline, which will be used to determine each participant's outcome. The scale is described as:
  1. Complete epithelialisation of the sentinel ulcer
  2. >50% reduction in sentinel ulcer surface area
  3. 20-50% reduction in sentinel ulcer surface area
  4. 0-20% reduction in sentinel ulcer surface area
  5. Any increase in sentinel ulcer surface area
  6. Development of new ulcers
  7. Amputation due to an ulcer
  8. All-cause death
Distribution of each of the individual components of the BCWAS, assessed at Weeks 4 | Week 4
  To determine whether addition of the intervention changes the distribution of each of the individual components of the BEAT-Calci Wound Assessment Scale, assessed at Weeks 4
  Scale described as:
  1. Complete epithelialisation of the sentinel ulcer
  2. >50% reduction in sentinel ulcer surface area
  3. 20-50% reduction in sentinel ulcer surface area
  4. 0-20% reduction in sentinel ulcer surface area
  5. Any increase in sentinel ulcer surface area
  6. Development of new ulcers
  7. Amputation due to an ulcer
  8. All-cause death
Distribution of each of the individual components of the BCWAS, assessed at Week 12 | Week 12
  To determine whether addition of the intervention changes the distribution of each of the individual components of the BEAT-Calci Wound Assessment Scale, assessed at Week 12
  Scale described as:
  1. Complete epithelialisation of the sentinel ulcer
  2. >50% reduction in sentinel ulcer surface area
  3. 20-50% reduction in sentinel ulcer surface area
  4. 0-20% reduction in sentinel ulcer surface area
  5. Any increase in sentinel ulcer surface area
  6. Development of new ulcers
  7. Amputation due to an ulcer
  8. All-cause death
Distribution of each of the individual components of the BCWAS, assessed at Week 26 | Week 26
  To determine whether addition of the intervention changes the distribution of each of the individual components of the BEAT-Calci Wound Assessment Scale, assessed at Week 26.
  Scale described as:
  1. Complete epithelialisation of the sentinel ulcer
  2. >50% reduction in sentinel ulcer surface area
  3. 20-50% reduction in sentinel ulcer surface area
  4. 0-20% reduction in sentinel ulcer surface area
  5. Any increase in sentinel ulcer surface area
  6. Development of new ulcers
  7. Amputation due to an ulcer
  8. All-cause death
Bates-Jensen Wound Assessment Tool - from Baseline to Week 4 | Week 4
  To determine whether addition of the intervention changes the severity of sentinel ulcer from Baseline, assessed at Week 4 using the Bates-Jensen Wound Assessment Tool
Bates-Jensen Wound Assessment Tool - from Baseline to Week 12 | Week 12
  To determine whether addition of the intervention changes the severity of sentinel ulcer from Baseline, assessed at Week 12, using the Bates-Jensen Wound Assessment Tool
Bates-Jensen Wound Assessment Tool - from Baseline to Week 26 | Week 26
  To determine whether addition of the intervention changes the severity of sentinel ulcer from Baseline, assessed at Week 26, using the Bates-Jensen Wound Assessment Tool
Sentinel ulcer surface area - from Baseline, assessed at Week 4 | Week 4
  To determine whether addition of the intervention changes the surface area of sentinel ulcer from Baseline, assessed at Week 4
Sentinel ulcer surface area - from Baseline, assessed at Week 12 | Week 12
  To determine whether addition of the intervention changes the surface area of sentinel ulcer from Baseline, assessed at Week 12
Sentinel ulcer surface area - from Baseline, assessed at Week 26 | Week 26
  To determine whether addition of the intervention changes the surface area of sentinel ulcer from Baseline, assessed at Week 26
All ulcers total surface area - from Baseline, assessed at Week 4 | Week 4
  To determine whether addition of the intervention changes the total surface area of all ulcers (not only the sentinel ulcer) from Baseline, assessed at Week 4
All ulcers total surface area - from Baseline, assessed at Week 12 | Week 12
  To determine whether addition of the intervention changes the total surface area of all ulcers (not only the sentinel ulcer) from Baseline, assessed at Week 12
All ulcers total surface area - from Baseline, assessed at Week 26 | Week 26
  To determine whether addition of the intervention changes the total surface area of all ulcers (not only the sentinel ulcer) from Baseline, assessed at Week 26
Change over time of self-reported pain | Week 26
  To determine whether addition of the intervention changes self-reported pain over time, assessed using the 0-to-10 Numerical Rating Scale
Self-reported pain at week 12 | Week 12
  To determine whether addition of the intervention changes self-reported pain use at week 12 assessed using the 0-to-10 Numerical Rating Scale
Change over time of analgesic use | Week 26
  To determine whether addition of the intervention changes analgesic use over time, as measured by cumulative weighted analgesia dose from baseline to week 26
Analgesic use week 12 | Week 12
  To determine whether addition of the intervention changes analgesic use over time, as measured by cumulative weighted analgesia dose from baseline to week 12
Composite self-reported pain and analgesic use over time | Week 26
  To determine whether addition of the intervention changes the composite outcome of self-reported pain (assessed using the 0-to-10 Numerical Rating Scale) and analgesic use over time
Composite self-reported pain and analgesic use at week 12 | Week 12
  To determine whether addition of the intervention changes the composite outcome of self-reported pain (assessed using the 0-to-10 Numerical Rating Scale) and analgesic use at week 12
Change in self-reported quality of life from Baseline to Week 4 | Week 4
  To determine whether addition of the intervention changes self-reported quality of life from Baseline, assessed at Week 4, using the EuroQoL EQ-5D-5L instrument
Change in self-reported quality of life from Baseline to Week 12 | Week 12
  To determine whether addition of the intervention changes self-reported quality of life from Baseline, assessed at Week 12, using the EuroQoL EQ-5D-5L instrument
Change in self-reported quality of life from Baseline to Week 26 | Week 26
  To determine whether addition of the intervention changes self-reported quality of life from Baseline, assessed at Week 26 using the EuroQoL EQ-5D-5L instrument
Time to first calciphylaxis-attributable infection from Baseline to Week 26 | Week 26
  Time in days to first calciphylaxis-attributable infection within 26 weeks post-randomisation
All-cause hospitalisation days | Weeks 0-26
  Count of all cause hospitalisation days (excluding day admissions for dialysis treatment within 26 weeks post-randomisation
Mortality | Up to 5 years
  Incidence of mortality, as derived from hospital reports, within 5-years post-randomisation
Kidney Transplantation | Up to 5 years
  Incidence of kidney transplantation, as derived from hospital reports, within 5-years post-randomisation
Calciphylaxis recurrence | Up to 5 years
  Incidence of calciphylaxis recurrence as derived from hospital reports, within 5-years post-randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Meg Jardine, Study Chair — University of Sydney
Locations (21):
- Australia (16):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast Hospital and Health Service, Birtinya, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Bundaberg Base Hospital, Bundaberg, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Townsville Hospital, Douglas, Queensland
  - Ipswich Hospital, Ipswich, Queensland
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Sunshine Hospital (Western Health), St Albans, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - Monash Medical Centre, Clayton
- New Zealand (5):
  - Dunedin Hospital, Dunedin
  - Auckland City Hospital (Auckland DHB), Grafton
  - North Shore Hospital (Waitemata DHB), Takapuna
  - Tauranga Hospital, Tauranga
  - Whangarei Hospital, Whangarei

IPD SHARING:
Plan to Share IPD: Yes
Trial data will be disseminated in the form of a publication to a relevant clinical journal and presentation at appropriate scientific conferences.
  Individual participant data that underlie the results reported, after de-identification (text, tables, figures, and appendices), may be shared with Investigators whose proposed use of the data has been approved by a review committee identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: To be confirmed
Access Criteria: * No data should be released that would compromise the trial, unless specifically for safety reasons.
  * There must be a strong scientific or other legitimate rationale for the data to be used for the requested purpose.
  * Investigators should have a period of exclusivity in which to pursue their aims with the data, before key trial data are made available to other researchers.
  * Adequate resources must be available in order to comply with the request, and the scientific aims of the study must justify the use of such resources.
  * Data release complies with the relevant regulations from all relevant countries.

REFERENCES:
- [Derived] Krishnasamy R, Jardine MJ; BEAT-Calci Trialists. Adaptive Designs for Clinical Trials in Nephrology. J Am Soc Nephrol. 2025 Jan 1;36(1):147-149. doi: 10.1681/ASN.0000000000000497. Epub 2024 Aug 26. No abstract available. PMID 39186385